CLINICAL TRIAL: NCT00709462
Title: A Phase I, Open-Label, Dose-Escalation, Multidose Study of CDX-1307, a Mannose Receptor-Targeted hCG-β Vaccine, in Patients With Incurable Breast, Colorectal, Pancreatic, Ovarian or Bladder Cancer (CDX-1307-01)
Brief Title: A Study of CDX-1307, in Patients With Incurable Breast, Colorectal, Pancreatic, Ovarian or Bladder Cancer (CDX 1307-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Celldex Therapeutics, Celldex Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX-1307-01
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Pancreatic Cancer; Bladder Cancer; Ovarian Cancer
Keywords: Breast cancer; Colorectal cancer; Pancreatic cancer; Bladder cancer; Ovarian cancer; Metastatic cancer; Locally advanced cancer; Cancer Vaccine; Vaccine
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis | interventions — CDX 1307

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: CDX1307

SUMMARY:
This research study is for individuals who have advanced breast, colon, pancreatic, ovarian or bladder cancer. Celldex Therapeutics, Inc. is testing a form of immune therapy (vaccine) to see if it can be used to make the immune system attack the cancer. The study includes administration of additional treatments, in combination, thought to enhance the immune response effect. (CDX 1307-01)

DETAILED DESCRIPTION:
Protocol CDX1307-01: CDX-1307 is an investigational drug that is being tested to see if it can stimulate the immune system (the cells and substances that protect the body from infection and foreign matter) of people with certain kinds of cancer. It is believed that the body's immune system can attack tumor cells and kill them. It is thought that immune cells recognize special proteins on the surface of tumors as a signal to fight the cancer. One of these proteins is called human chorionic gonadotropin-beta (hCG-β) and is found on several types of cancers including breast, colorectal, pancreatic, bladder and ovarian. The study drug will be given as an injection under the skin (an intradermal or intracutaneous injection). In addition, the study includes combination with TLR agonists, which are thought to stimulate the immune response against tumor cells.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have read, understood, and provided written informed consent and HIPAA authorization after the nature of the study has been fully explained.
2. Patients must be 18 years of age or older.
3. Patients with incurable breast, colorectal, pancreatic, ovarian or bladder cancer with measurable or evaluable disease.
4. Patients who have never received prior hCG-β therapy.
5. Patients for whom therapy with potential survival benefit is available, or disease-specific palliation is the goal of therapy, must have received these appropriate standard of care therapies and experienced recurrence or progression while on that care. If no such therapy is available, patients with progressive disease may be enrolled. Patients who have refused standard of care options known to provide potential survival benefit or disease specific palliation are not eligible for this study.
6. At least 4 weeks must have elapsed between prior therapy and first dose of the vaccine. Prior radiation therapy must be completed at least 4 weeks prior to the first vaccine dose. No prior radiopharmaceuticals within 8 weeks prior to the first vaccine dose. The patient must have recovered from any clinically significant toxicity experienced during prior treatment(s).
7. Patients on the following medications may be enrolled into the study if the medications were initiated 4 weeks or longer prior to screening and if no dosing changes are anticipated during the study.

   1. Hormonal therapy including gonadotropin releasing hormone (GnRh) agonist, antiandrogens, selective estrogen receptor modulators (SERMs), aromatase inhibitors, and progestins.
   2. Bisphosphonates.
8. Patients must have an ECOG Status of 0 or 1.
9. Patients must have a life expectancy ≥ 16 weeks.
10. Male patients who are sexually active must agree to practice an effective form of barrier contraception during the course of the study.
11. Screening laboratory values must meet the following criteria:

    * Neutrophils ≥1.5 x109/L
    * Platelets >100 x109/L
    * Hemoglobin <10 g/dL
    * Creatinine <2 mg/dL
    * AST <2 X ULN
    * Bilirubin <2 X ULN unless due to Gilbert's syndrome upper limit of normal.

Laboratory abnormalities attributed to liver involvement with cancer but outside of the normal range will be allowed if they do not exceed the following limits:

* AST <4 X ULN
* Bilirubin <4 X ULN

Exclusion Criteria

1. Since treatment with CDX-1307 theoretically may cause permanent sterility, women of childbearing potential will be excluded (women who participate in this study must be post-menopausal [absence of menses for at least 1 year] and/or surgically incapable of bearing children).
2. Previous administration of hCG-β vaccine or therapy.
3. Concurrent treatment with immunosuppressive or immunomodulatory agents.
4. Positive tests for HIV, HBV or HCV.
5. Patients with an active systemic infection requiring antibiotic treatment or a fever over 100°F within 72 hours prior to enrollment.
6. Generalized dermatologic conditions (such as allergic reactions, infection, edema, or scarring) that will not allow easy access for study drug administration or evaluation of localized adverse events.
7. Patients with active central nervous system metastases, unless previously treated and asymptomatic for 2 months and not progressive in size or number for 2 months.
8. History of a second malignancy, except for adequately treated and cured basal or squamous cell skin cancer or any other cancer from which the patient has been disease-free for ≥ 5 years.
9. History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, or known hypersensitivity to GM-CSF, or yeast derived products.
10. Patients with any of the following conditions: myocardial infarction within 1 year of screening, congestive heart failure (unless LVEF ≥ 50% as determined by MUGA within 30 days of screening), uncontrolled hypertension (≥ 160 mm Hg/systolic and ≥ 100 mm Hg/diastolic), symptomatic or life-threatening arrhythmia persistent on medication at screening, or clinically evident chronic lung disease unless lung capacity ≥ 55% or FEV1 ≥ 60% at screening.
11. Any underlying medical condition that in the Principal Investigator's opinion will make the administration of study drug hazardous to the patient or would obscure the interpretation of adverse events.
12. Medical condition requiring the use of systemic corticosteroids (must be discontinued at least 4 weeks prior to enrollment. The use of inhaled corticosteroids is acceptable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2004-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To establish the safety and tolerability profile of CDX-1307 in patients with incurable breast, colorectal, pancreatic, ovarian or bladder cancer, alone and in combination with adjuvants. | up to 2 years or until progression

SECONDARY OUTCOMES:
To evaluate dose-limiting toxicities, immune response, and clinical activity (tumor response and time to progression) | up to 2 years or until progression

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Duke University, Durham, North Carolina
  - Carolina BioOncology Institute Cancer, Huntersville, North Carolina